CLINICAL TRIAL: NCT02709395
Title: Evaluation of a Novel Electronic Transanal Irrigation System - Navina™ Smart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NAV-0003
Record Dates: First submitted 2016-02-25; First posted 2016-03-16 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-04

CONDITIONS: Neurogenic Bowel
MeSH Terms: conditions — Neurogenic Bowel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Navina Smart (Experimental): Navina Smart will be used, during 4 weeks, for transanal irrigation (TAI).
  Interventions: Device: Navina Smart

INTERVENTIONS:
Device: Navina Smart — Transanal irrigation at the same frequency as subject used before enrollment.

SUMMARY:
This study is designed as an open, prospective, single arm, multicenter study in order to investigate patient satisfaction, perception and compliance for the novel Navina Smart, a transanal irrigation (TAI) system. Approximately 30 male and female subjects who are currently practicing TAI, will be followed during a 4-week period of use of Navina Smart. Observational data on satisfaction, perception, compliance, bowel regimen, TAI therapy and TAI frequency will be collected via patient reported outcome (PRO) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Males and females, aged 18 years and over
3. Practice TAI since at least 2 months and at least two times per week
4. Able to read and fill out a paper PRO questionnaire as judged by the principal investigator or a sub-investigator

Exclusion Criteria:

1. Any confirmed or suspected diagnosis of anal or rectal stenosis, active inflammatory bowel disease, acute diverticulitis, severe diverticulosis, colorectal cancer, ischemic colitis, history of life-threatening autonomic dysreflexia, bleeding disorders, unspecified peri-anal conditions
2. Untreated rectal impaction
3. Any radiotherapy to the pelvis
4. Any current treatment with anticoagulants (not including aspirin or clopidogrel)
5. Any current treatment with long-term systemic steroid medication (not including inhalation agents and/ or local topical treatment)
6. Any prior rectal or colonic surgery (not including anal procedures >3 months ago, e.g. haemorrhoid excision)
7. Anal, rectal and/or colonic endoscopic polypectomy within the previous 4 weeks
8. Overt or planned pregnancy
9. Ongoing symptomatic urinary tract infection as judged by the principal investigator or a sub-investigator
10. Diagnosed psychiatric illness, considered as unstable by the principal investigator or a sub-investigator
11. Involvement in the planning and conduct of the study (applies to both Wellspect HealthCare staff and staff at the study site)
12. Previous enrolment in the present study
13. Participation in another clinical study within the last 30 days that may interfere with the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Neurologiska kliniken, Karolinska Universitetssjukhuset Solna, Stockholm, Sweden
- Gastrointestinal Physiology Unit, University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Navina Smart
Started | 28 (28 subjects enrolled and found to be eligible for further study participation after screening.)
Completed | 19
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Navina Smart
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 53.17 [24.06 to 72.79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Bowel Management at Baseline - Satisfaction [Count of Participants; unit: Participants] — The Baseline Questionnaire is a study-specific, non-validated instrument, developed by Wellspect HealthCare. The Baseline Questionnaire is self-administered and was completed by the subjects at Visit 1.
  Participants
    Not Satisfied - Not satisfied at all | 11
    Neutral | 7
    Satisfied - Completely satisfied | 10
TAI therapy at Baseline [Count of Participants; unit: Participants] — The Baseline Questionnaire is a study-specific, non-validated instrument, developed by Wellspect HealthCare. The Baseline Questionnaire is self-administered and was completed by the subjects at Visit 1.
  Participants
    Peristeen | 28
    Other | 0
Time spent bowel management at Baseline [Mean (Full Range); unit: minutes] — Measure Description: The Baseline Questionnaire is a study-specific, non-validated instrument, developed by Wellspect HealthCare. The Baseline Questionnaire is self-administered and was completed by the subjects at Visit 1. Population: Data missing for 4 subjects, no response received
  minutes
    number analyzed (Participants) | 24
    (all) | 54.90 [0 to 270]

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire Measuring Subjects' Satisfaction of Navina Smart
Description: PRO Questionnaire, completed by each subject after 4 weeks of using Navina Smart, collecting data on subject's assessment of satisfaction when using the study device.
  Satisfaction was assessed in a range of ways through different questions to be answered by each subject. For example each subject received the question "If possible, would you consider continuing using the Navina Smart system?"
Time Frame: 4 weeks
Population: Intention To Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Navina Smart
Number analyzed (Participants) | 28
Participants
  Answer missing | 1
  Yes | 14
  No | 13

2. Primary Outcome: Questionnaire Measuring Subjects' Perception of Navina Smart
Description: PRO Questionnaire, completed by each subject after 4 weeks of using Navina Smart, collecting data on subject's assessment of perception when using the study device.
  For example, each subject answered the following question regarding perception: "How satisfied are you with the Navina Smart System?"
Time Frame: 4 weeks
Population: Intention To Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Navina Smart
Number analyzed (Participants) | 28
Participants
  Answer missing | 1
  Neutral, satisfied or very satisfied with Navina | 18
  Not satisfied with Navina | 9

3. Primary Outcome: Questionnaire Measuring Subjects' Compliance of Navina Smart
Description: PRO Questionnaire, completed by each subject after 4 weeks of using Navina Smart, collecting data on subject's compliance towards the study device.
  For example, each subject answered the following question "Did you use the Navina Smart system for 4 weeks?"
Time Frame: 4 weeks
Population: Intention To Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Navina Smart
Number analyzed (Participants) | 28
Participants
  Answer missing | 0
  Yes | 19
  No | 9

4. Secondary Outcome: Adverse Events (AEs), Adverse Device Effects (ADEs), Serious Adverse Events (SAEs) Related to Navina Smart
Description: Total numbers and types of AEs, ADEs and SAEs observed by the study staff or spontaneously reported from the patient.
Time Frame: 4 weeks
Population: Safety Analysis Set
Measure: Number; unit: number of events
Arm/Group | Navina Smart
Number analyzed (Participants) | 28
number of events | 3

ADVERSE EVENTS:
Time Frame: The safety of Navina Smart, e.g. registration of Adverse Events (AEs), Adverse Device Effects (ADEs), Serious Adverse Events (SAEs), were collected throughout the study period for 4 weeks of each participating subject.
Arm/Group | Navina Smart
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 3/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Navina Smart (N=28)
Broke left leg (Injury, poisoning and procedural complications) | 1
Vomiting (Gastrointestinal disorders) | 1
Skin infection elbow (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes